CLINICAL TRIAL: NCT07358715
Title: A Multimodal Liquid Biopsy-Based Assay as a Pre-Screening Test Before Low Dose CT Thorax (LDCT) to Streamline Lung Cancer Screening in High-Risk Individuals
Brief Title: Liquid Biopsy-Based Pre-Screening to Streamline LDCT Lung Cancer Screening in High-Risk Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Gene Solutions (Industry)
Responsible Party: Principal Investigator, Haematology-Oncology, Prof. Lee Soo Chin, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 2024-3143
Record Dates: First submitted 2026-01-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Lung Neoplasms; Early Lung Cancer Detection; Cancer Screening; High-Risk Populations
Keywords: Liquid biopsy; DNA methylation; Exosomes; Blood-based screening; Low-dose CT; LDCT; Lung cancer screening; Early cancer detection; High-risk individuals; Never-smokers; Multimodal assay
MeSH Terms: conditions — Lung Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to protocol-defined diagnostic procedures based on cohort classification (high-risk individuals without lung cancer, early-stage lung cancer patients, or advanced-stage lung cancer patients). High-risk participants undergo liquid biopsy testing followed by LDCT screening, with CT-PET performed if liquid biopsy results are positive and LDCT findings are negative. Cancer cohorts undergo liquid biopsy testing only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Risk Individuals Without Known Lung Cancer (Experimental): High-risk individuals without a prior diagnosis of lung cancer undergo blood-based liquid biopsy testing followed by low-dose CT (LDCT) thorax screening as per the study protocol. Participants with positive liquid biopsy results and negative LDCT findings will be offered a study-funded CT-PET scan for further evaluation.
  Interventions: Diagnostic Test: Liquid Biopsy (SPOT-MAS Assay); Diagnostic Test: Exosome-Based Liquid Biopsy Assay; Diagnostic Test: Low-Dose CT Thorax (LDCT)
- Early-Stage Lung Cancer Patients (Stage I-II) (Experimental): Participants with histologically confirmed early-stage lung cancer (Stage I-II) undergo blood collection for liquid biopsy testing to evaluate assay performance in early disease.
  Interventions: Diagnostic Test: Liquid Biopsy (SPOT-MAS Assay); Diagnostic Test: Exosome-Based Liquid Biopsy Assay
- Advanced-Stage Lung Cancer Patients (Stage III-IV) (Experimental): Participants with histologically confirmed advanced-stage lung cancer (Stage III-IV) undergo blood collection for liquid biopsy testing to evaluate assay performance in advanced disease.
  Interventions: Diagnostic Test: Liquid Biopsy (SPOT-MAS Assay); Diagnostic Test: Exosome-Based Liquid Biopsy Assay

INTERVENTIONS:
Diagnostic Test: Liquid Biopsy (SPOT-MAS Assay) — Blood-based genome-wide DNA methylation assay performed on plasma samples to detect tumor-associated methylation patterns suggestive of lung cancer.
Diagnostic Test: Exosome-Based Liquid Biopsy Assay — Blood-based assay analyzing exosome-associated biomarkers to support early detection of lung cancer.
Diagnostic Test: Low-Dose CT Thorax (LDCT) — Low-dose computed tomography of the thorax performed for lung cancer screening
  Arms: High-Risk Individuals Without Known Lung Cancer

SUMMARY:
This study evaluates the feasibility and cost-effectiveness of using a blood-based liquid biopsy assay as a pre-screening tool before low-dose CT (LDCT) for lung cancer screening. By identifying individuals unlikely to have lung cancer, this approach aims to reduce unnecessary LDCT scans, radiation exposure, and healthcare costs, while improving early detection, particularly among high-risk individuals including never-smokers with a family history of lung cancer.

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related mortality worldwide, largely due to late-stage diagnosis. Low-dose computed tomography (LDCT) has been shown to reduce lung cancer mortality in high-risk populations; however, its population-level implementation is limited by high false-positive rates, radiation exposure, cost, and poor uptake. These challenges are particularly relevant in Asian populations, where a substantial proportion of lung cancer occurs among never-smokers, for whom optimal screening strategies remain unclear.

Recent advances in liquid biopsy technologies have enabled the detection of circulating tumor-derived signals, including DNA methylation patterns and extracellular vesicle-associated biomarkers, offering a minimally invasive approach for early cancer detection. Multimodal liquid biopsy assays may serve as an effective pre-screening tool to identify individuals who are unlikely to have lung cancer and who may not require immediate LDCT screening.

This prospective, interventional study aims to evaluate the feasibility, diagnostic performance, and potential cost-effectiveness of a multimodal liquid biopsy-based assay as a pre-screening strategy prior to LDCT for lung cancer screening in high-risk individuals. The study includes three cohorts: (1) Healthy but high-risk individuals, without a prior diagnosis of lung cancer, (2) patients with early-stage lung cancer (Stage I-II), and (3) patients with advanced-stage lung cancer (Stage III-IV).

Healthy, but high-risk individuals will undergo blood collection for two liquid biopsy assays: a genome-wide DNA methylation-based assay (SPOT-MAS) and an exosome-based biomarker assay. All healthy individuals will subsequently undergo LDCT thorax screening. In cases where the SPOT-MAS result is positive but LDCT findings are negative, participants will be offered a study-funded CT-PET scan, within 3 months of blood collection to further evaluate the presence of malignancy. If CT-PET is negative, participants will be referred for further follow-up tests, e.g., Oesophago-Gastro-Duodenoscopy (OGD) / colonoscopy/ mammogram (funded by the study) or no further tests, at physician's discretion. Healthy, high-risk volunteers with positive LDCT results will be referred to a respiratory physician for further evaluation as per routine clinical pathway (not funded by the study). Healthy, high-risk individials who are negative on both tests will have no further study-mandated visits. In rare cases where the SPOT-MAS result is inconclusive, a second blood sample (10 mL) will be collected after 1month but within 6 months after the first blood draw.

Early- and advanced-stage lung cancer patients will undergo blood collection for liquid biopsy testing only, to assess assay performance across different disease stages.

The primary outcomes include the negative predictive value of the liquid biopsy assays and the proportion of high-risk individuals who could potentially be spared LDCT screening based on negative liquid biopsy results. Secondary outcomes include the sensitivity, specificity, and predictive values of the assays compared with imaging and clinical diagnosis, as well as exploratory analyses of the cost-effectiveness of a liquid biopsy-guided screening strategy.

By evaluating a blood-based pre-screening approach integrated with imaging, this study aims to inform more efficient and personalized lung cancer screening strategies that may reduce unnecessary imaging, radiation exposure, and healthcare costs, while maintaining early detection performance in high-risk populations.

ELIGIBILITY:
Inclusion Criteria

High-Risk Individuals (n = 100)

* No prior history of lung cancer
* Meets one of the following high-risk definitions:

  * Current or former smoker (quit within the past 15 years), aged 55-74 years, with a smoking history of ≥30 pack-years; OR
  * Never-smoker aged 55-75 years with a first-degree family history of lung cancer
* Able and willing to provide written informed consent

Early-Stage Lung Cancer Patients (n = 20)

* Aged ≥21 years
* Histologically or clinically confirmed stage I-II lung cancer
* Treatment-naïve (no prior surgery, chemotherapy, radiotherapy, or immunotherapy for lung cancer)
* Able and willing to provide written informed consent

Advanced-Stage Lung Cancer Patients (n = 20)

* Aged ≥21 years
* Histologically or clinically confirmed stage III-IV lung cancer
* Treatment-naïve (no prior systemic or local therapy for lung cancer)
* Able and willing to provide written informed consent

Exclusion Criteria

Applicable to All Participants

* Pregnant or breastfeeding women
* Inability or unwillingness to comply with study procedures

High-Risk Individuals Only

* Known allergy or contraindication to CT contrast agents
* Prior low-dose CT (LDCT), CT thorax, or PET-CT performed within 12 months prior to enrollment

Lung Cancer Cohorts Only

• Receipt of any prior cancer-directed treatment for lung cancer

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative Predictive Value of Liquid Biopsy Pre-Screening | 12 months
  Description:
  Negative predictive value of the liquid biopsy assay (SPOT-MAS), defined as the proportion of participants with a negative liquid biopsy result who have no lung cancer detected by low-dose computed tomography (LDCT) and clinical follow-up.
  Unit of Measure: Proportion (%)
Reduction in Unnecessary LDCT Screening | 12 months
  Proportion of high-risk participants who receive a negative liquid biopsy (SPOTMAS) result, representing individuals who may be eligible to defer LDCT screening under a liquid biopsy-guided pre-screening strategy.
  Unit of Measure: Proportion (%)

SECONDARY OUTCOMES:
Diagnostic Accuracy of Liquid Biopsy Assays | 12 months
  Sensitivity, specificity and positive predictive value of liquid biopsy assays (SPOT-MAS and exosome-based assays) compared with LDCT and clinical follow-up.
  Unit of Measure: Proportion (%)
Cost-Effectiveness of Liquid Biopsy Pre-Screening | 12 months
  Comparative cost analysis (Mean total screening-related cost) of liquid biopsy-guided screening versus LDCT-only screening.
  Unit of Measure: Cost (USD per participant)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No